CLINICAL TRIAL: NCT02975063
Title: Alive & Thrive Nigeria Impact Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: FHI 360 (Other); University of North Carolina, Chapel Hill (Other); TNS RMS Nigeria, Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08100206
Record Dates: First submitted 2016-10-19; First posted 2016-11-29 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2020-08

CONDITIONS: Complementary Feeding
Keywords: Exclusive breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A&T IYCF intervention (Experimental): A&T IYCF intervention is includes comprehensive IYCF counseling which includes intensive activity that aims to deliver one-on-one counseling at home or in a health facility.
  Interventions: Behavioral: A&T IYCF intervention
- Control (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: A&T IYCF intervention — (1) Interpersonal communication through frontline workers/volunteers to increase mothers' knowledge and practice of optimal infant and young child feeding (IYCF) behaviors. Interpersonal communication will involve multiple contacts with mothers and an array of IYCF messages; (2) Community mobilization activities to raise awareness of the benefits of optimal IYCF practices among opinion leaders and family members, and increase their support to mother for IYCF; (3) Training of facility and community-based health workers on IYCF to improve their ability to support mothers and provide timely information on IYCF; and (4) Mass media communication on IYCF.
  Arms: A&T IYCF intervention

SUMMARY:
Investigators will use a cluster-randomized design to evaluate the overall impact of the Alive & Thrive infant and young child feeding communication strategies in Lagos and Kaduna States, Nigeria. The impact in each state and in a subset of urban local government areas (LGAs) will also be tested.This is a mixed methods evaluation; the quantitative data will be complemented by qualitative data obtained from different groups targeted by or involved in the program.

DETAILED DESCRIPTION:
Adequate nutrition during the first 1,000 days is necessary for children to grow and develop to their full potential. Alive & Thrive (A&T) contributes to better nutrition during the first 1,000 days by promoting improved infant and young child feeding (IYCF) practices. A&T is expanding its efforts to Nigeria and will target Lagos and Kaduna States. In Nigeria, 33% of infants are breastfed within 1 hour of delivery, 60% are given other fluids in the first 3 days of life, and only 17% of children 0-5.9 months are exclusively breastfed. Approximately 60% of children 6 to 23 months achieve the minimum meal frequency for their age and 19% are fed four or more food groups per day. To address these gaps in optimal IYCF practices, A&T will use an implementation framework for IYCF impact at scale that includes advocacy, interpersonal communication and community mobilization, mass communication, and strategic use of data. The A&T intervention will be compared to mass media communication on IYCF, which will be provided throughout the two states. LGAs in Lagos and Kaduna will be randomly allocated such that two-thirds receive the A&T intervention and one-third are assigned to the comparison group. The primary objectives of the evaluation are to measure the impact of the A&T intervention on IYCF practices among mothers with children 0-23 months of age overall, in each state, and in a subset of urban LGAs. Secondary evaluation objectives are to document: the type, quantity, and timing of the implementation of A&T program activities; coverage levels A&T achieves with different program activities; extent to which A&T increases knowledge and awareness of optimal IYCF practices among women with children 0 to 23 months and health providers; extent to which A&T improves the capacity of health providers to counsel mothers on IYCF; and extent to which A&T improves the capacity of stakeholders to implement community-based activities that support optimal IYCF practices.

ELIGIBILITY:
Inclusion Criteria:

* For mother's survey:
* Women of reproductive age (15-49 years),
* Must be married if 15-17 years,
* Has a child 0-23 months
* For provider's survey:
* Male or female,
* 18 years or older
* Works in a government or private health facility or works as a community pharmacist, private patent medicine vendor, or traditional birth attendant

Exclusion Criteria:

-

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15169 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding on the day preceding the interview. | 2 years
  The proportion of infants 0-5 months who were exclusively breastfed on the previous day.

SECONDARY OUTCOMES:
Exclusive breastfeeding from 0-5 months. | 2 years
  The proportion of children who were exclusively breastfed from 0-5 months.
Breastfeeding within 1 hour of birth. | 2 years
  The proportion of children 0-23 months who were breastfed within 1 hour of birth.
Minimum dietary diversity. | 2 years
  The proportion of children 6-23 months who were fed the minimum number of food groups on the previous day based on the WHO infant and young child feeding guidelines.
Minimum meal frequency. | 2 years
  Description: The proportion of children 6-23 months who were fed the minimum number of meals on the previous day based on the World Health Organization infant and young child feeding guidelines.
Mothers' accurate knowledge of optimal infant and young child feeding practices. | 2 years
  Mothers' accurate knowledge of:
  * Optimal timing of breastfeeding initiation
  * Optimal duration of exclusive breastfeeding
  * Solution to common breastfeeding problems
  * Optimal timing to introduce complementary foods
  * Optimal dietary diversity and frequency of complementary feeding from 6-23 months
Health providers' knowledge of optimal infant and young child feeding practices. | 2 years
  Providers' accurate knowledge of:
  * Optimal timing of breastfeeding initiation
  * Optimal duration of exclusive breastfeeding
  * Solution to common breastfeeding problems
  * Optimal timing to introduce complementary foods
  * Optimal dietary diversity and frequency of complementary feeding from 6-23 months

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flax, Principal Investigator — RTI International; Mariam Fagbemi, Principal Investigator — TNS RMS Nigeria, Ltd.
Locations (2):
- Nigeria (2):
  - Kantar TNS RMS, Ikeja, Lagos
  - Kantar TNS RMS, Kaduna

REFERENCES:
- [Derived] Flax VL, Fagbemi M, Schnefke CH, Kawu AA, Edwards S, Unangst J, Bose S. Impacts of a social and behavior change communication program implemented at scale on infant and young feeding practices in Nigeria: Results of a cluster-randomized evaluation. PLoS One. 2022 Dec 8;17(12):e0277137. doi: 10.1371/journal.pone.0277137. eCollection 2022. PMID 36480569